CLINICAL TRIAL: NCT03873675
Title: Trends in Parathyroid Hormone Plasma Concentration in Multi-organ Failure Critically Ill Patients Undergoing Regional Citrate Anticoagulation Continuous Renal Replacement Therapies - Prospective Observational Study.
Brief Title: Parathyroid Hormone Kinetics During CRRT
Status: Completed | Type: Observational
Sponsor: Uniwersytecki Szpital Kliniczny w Opolu (Other)
Responsible Party: Principal Investigator, Tomasz Czarnik, MD PhD, Principal Investigator, Uniwersytecki Szpital Kliniczny w Opolu
Other Study IDs: AKIparathormoneCRRTstudy
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Critical Illness; Multi Organ Failure; Renal Failure; Circulatory Failure; Respiratory Failure
Keywords: acute kidney injury; parathyroid hormone; continuous renal replacement therapy; citrate anticoagulation; intensive care
MeSH Terms: conditions — Critical Illness; Multiple Organ Failure; Renal Insufficiency; Shock; Respiratory Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples (10-20ml) taken from the arterial catheter every 12 hours
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Multi-organ failure with acute kidney injury critically ill patients admitted to the intensive care unit undergoing regional citrate anticoagulation continuous renal replacement therapy by means of continuous veno-venous hemodiafiltration (CVVHDF). Multi-organ failure is defined as a respiratory, circulatory and renal failure.
  Interventions: Diagnostic Test: parathyroid hormone

INTERVENTIONS:
Diagnostic Test: parathyroid hormone — 10-20ml blood samples taken from the arterial catheter every 12 hours to obtain parathyroid hormone serum concentration. 6-8 samples per patient

SUMMARY:
The objective of this study is to assess the parathyroid hormone serum concentrations and kinetics in critically ill patients admitted to the intensive care unit due to multi-organ failure and undergoing citrate anticoagulation continuous renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory failure
* Acute circulatory failure
* acute kidney injury treated with regional citrate anticoagulation continuous renal replacement therapy by means of continuous veno-venous hemodiafiltration (CVVHDF
* continuous renal replacement therapy started no later than 48 hours after admission
* SOFA score 5 or more

Exclusion Criteria:

* age less than 18 years
* acute liver failure
* hypercalcemia at admission (total calcium plasma level > 10.6 mg/dL; total ionized calcium plasma level > 1.35 mmol/L
* parathyroid glands disease
* end stage renal disease
* therapeutic plasma exchange
* extracorporeal membrane oxygenation
* unfavorable outcome (death) predicted within 72 hours (as assessed by investigator)
* lack of relatives consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multi-organ failure with acute kidney injury critically ill patients admitted to the critical care unit undergoing regional citrate anticoagulation continuous renal replacement therapy by means of continuous veno-venous hemodiafiltration (CVVHDF). Multi-organ failure is defined as a respiratory, circulatory and renal failure.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
The change in parathyroid hormone serum concentration during regional citrate anticoagulation continuous renal replacement therapy (CRRT) in the acute phase of critical illness. | 96 hours
  The first parathyroid hormone serum level will be measured before the start of CRRT (the zero point) Next measurements will be performed every 12 hours. Minimal number of measurements - 6, maximal - 8 per patient.

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (3):
  - Department of Endocrinology, Diabetology and Isotope Therapy, Wroclaw Medical University, Poland., Wroclaw, Lower Silesian Voivodeship
  - Department of Endocrinology, Szpital Wojewodzki w Opolu, Opole, Silesian Voivodeship
  - Department of Anesthesiology and Intensive Care, Uniwersytecki Szpital Kliniczny w Opolu, Opole, Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Czarnik A, Gawda R, Piwoda M, Marszalski M, Molsa M, Pietka M, Bolanowski M, Czarnik T. Parathyroid hormone serum concentration kinetic profile in critically ill patients undergoing continuous renal replacement therapies: a prospective observational study. Endokrynol Pol. 2021;72(4):329-335. doi: 10.5603/EP.a2021.0034. Epub 2021 May 19. PMID 34010434